CLINICAL TRIAL: NCT06611891
Title: Evaluation of Somatostatin Receptor Expression in PET 68Ga-DOTATOC in Patients Followed for Metastatic Breast Cancer
Acronym: DOTABREAST
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC21.0432
Record Dates: First submitted 2023-04-20; First posted 2024-09-25 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Metastatic
Keywords: Breast Cancer Metastatic; Somatostatin Receptor Expression; PET-SCAN; 68Ga-DOTATOC; Nuclear Oncology; 177-Lu-Oxodotreotide; DOTATOC
MeSH Terms: interventions — Ga(III)-DOTATOC

STUDY DESIGN:
Intervention Model Description: 25 patients: 25 patients with breast cancer labeled on the primary lesion ER+HER2-
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Performing a 68Ga-Dotatoc PET scan in patients followed for metastatic breast cancer. (Experimental): 1. Prescreening of the patient followed for metastatic breast cancer during the routine care
  2. V1 Selection: Patient's selection in the Nuclear Medicin or Oncology department
  3. V2 Inclusion: The day of the 68Ga-Dotatoc PET scan in the Nuclear Medicin department
  4. V3 End of study visit, the same day after the 68Ga-Dotatoc PET scan.
  Interventions: Drug: 68Ga-DOTATOC

INTERVENTIONS:
Drug: 68Ga-DOTATOC — Slow direct intravenous injection

SUMMARY:
DOTABREAST: Evaluation of Somatostatin Receptor Expression in PET 68Ga-DOTATOC in Patients Followed for Metastatic Breast Cancer

This is a prospective, monocentric, non-controlled, non-randomized, open-label, interventional study.

DETAILED DESCRIPTION:
In women, breast cancer is the 1st largest cancer and accounted for 31% of new cancer cases in women in 2017. With 11,913 deaths in 2015, breast cancer is the 1st largest cancer death in women (19%) and the 3rd largest cancer death (men and women included) after lung and colorectal cancer. At initial diagnosis at any stage, approximately 31% of patients have regional lymph node involvement and 5 to 10% present metastatic involvement from the outset. Progression to a metastatic form occurs in about 20% of cases. The risk of metastatic evolution is variable depending on the histological subtype and is a major prognostic event directly impacting overall survival. DOTATOC-68Ga PET scans allows in vivo evaluation of SST2 somatostatin receptor expression. Its use is widely validated in clinical practice for the assessment of extension of neuroendocrine tumors. It is also being used to evaluate the feasibility of SST2-targeted internal radiotherapy therapy with Lutathera (177Lu-Oxodotreotide) in patients with metastatic small intestine neuroendocrine tumours.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Patients with metastatic breast cancer who have completed at least one first line of systemic therapy for metastatic breast cancer
* Patient labeled on the primary lesion ER+HER2- (20)
* Presence of metastatic liver and bone lesions identifiable with 18F-FDG PET-Scan
* Presence of at least 10 identifiable secondary lesions in 18F-FDG PET-Scan
* No therapeutic change between 18F-FDG PET-Scan and 68Ga-DOTATOC PET-Scan.
* Performing the PET scan with 68Ga-DOTATOC within a maximum of 21 days after the 18F-FDG PET-Scan
* Person affiliated to or benefiting from social security
* Person who has given written informed consent

Exclusion Criteria:

* Patients followed or with history of other active neoplastic pathology (including neuroendocrine tumor)
* Known allergy to 68Ga-DOTATOC or its excipients
* Subject refusing to sign the consent to participate
* Minor subject
* Subject excluded from another study
* Persons referred to Articles L1121-5 to L1121-8 of the Public Health Code (CSP)
* Subject cannot be contacted in case of emergency

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Presence of lesions expressing SST2 receptors in 68Ga-DOTATOC in patients followed for metastatic breast cancer | Baseline (during the PET examination)
  Krenning Score >2

SECONDARY OUTCOMES:
Distribution of SST2 receptor overexpression by 68Ga-DOTATOC PET compared to 18F-FDG PET lesions. | Baseline (during the PET examination)
  Lesion-by-lesion analysis of lesion fixation intensity on 68Ga-DOTATOC PET (Krenning score (requires comparison to the liver and spleen (or kidney if not applicable) and calculated between 0 and 4) and PET quantification parameters).
Disease proportion with SST2 receptor overexpression by 68Ga-DOTATOC PET compared to known metastatic disease by 18F-FDG PET | Baseline (during the PET examination)
  Disease volume per patient with overexpression of SST2 receptors in 68Ga-DOTATOC PET compared to metabolic volume in 18F-FDG PET
Expression of SST2 receptors of lesions as a function of different metastatic sites, via the Krenning score | Baseline (during the PET examination)
  Krenning Score (from 0 to 4, 0 is none and 4 is greater than that of spleen, lesion with very low or no DOTATOC uptake (Score 0 or 1) are consider as a negative lesion, lesion with DOTATOC uptake ≥ 2 are consider as a positive lesion)
Expression of SST2 receptors of lesions as a function of different metastatic sites, via the PET quantification parameters. | Baseline (during the PET examination)
  PET quantification parameters (SUV max and SUV mean)
Correlation between the metabolic activity of 18F-FDG PET lesions and the expression of SST2 receptors in 68Ga-DOTATOC PET per lesion and per patient. | Baseline (during the PET examination)
  Comparison between 68Ga-DOTATOC PET and 18F-FDG PET (Krenning score and PET quantification parameter) per lesion and per patient.
Clinica predictors of overexpression of SST2 receptors in 68Ga-DOTATOC PET per patient | Baseline (during the PET examination)
  Clinical data prior to PET at 68Ga-DOTATOC per patient
Biological predictors of overexpression of SST2 receptors in 68Ga-DOTATOC PET per patient | Baseline (during the PET examination)
  Biological data prior to PET at 68Ga-DOTATOC per patient
Histological predictors of overexpression of SST2 receptors in 68Ga-DOTATOC PET per patient | Baseline (during the PET examination)
  Histological data prior to PET at 68Ga-DOTATOC per patient
Imaging predictors of overexpression of SST2 receptors in 68Ga-DOTATOC PET per patient | Baseline (during the PET examination)
  Imaging data prior to PET at 68Ga-DOTATOC per patient
Clinical predictors of overexpression of SST2 receptors in 68Ga-DOTATOC PET by lesion | Baseline (during the PET examination)
  Clinical data prior to PET at 68Ga-DOTATOC per lesion
Biological predictors of overexpression of SST2 receptors in 68Ga-DOTATOC PET by lesion | Baseline (during the PET examination)
  Biological data prior to PET at 68Ga-DOTATOC per lesion
Histological predictors of overexpression of SST2 receptors in 68Ga-DOTATOC PET by lesion | Baseline (during the PET examination)
  Histological data prior to PET at 68Ga-DOTATOC per lesion
Imaging predictors of overexpression of SST2 receptors in 68Ga-DOTATOC PET by lesion | Baseline (during the PET examination)
  Imaging data prior to PET at 68Ga-DOTATOC per lesion

CONTACTS AND LOCATIONS:
Overall Officials: Loic DJAILEB, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strosberg J, El-Haddad G, Wolin E, Hendifar A, Yao J, Chasen B, Mittra E, Kunz PL, Kulke MH, Jacene H, Bushnell D, O'Dorisio TM, Baum RP, Kulkarni HR, Caplin M, Lebtahi R, Hobday T, Delpassand E, Van Cutsem E, Benson A, Srirajaskanthan R, Pavel M, Mora J, Berlin J, Grande E, Reed N, Seregni E, Oberg K, Lopera Sierra M, Santoro P, Thevenet T, Erion JL, Ruszniewski P, Kwekkeboom D, Krenning E; NETTER-1 Trial Investigators. Phase 3 Trial of 177Lu-Dotatate for Midgut Neuroendocrine Tumors. N Engl J Med. 2017 Jan 12;376(2):125-135. doi: 10.1056/NEJMoa1607427. PMID 28076709
- [Background] Frati A, Rouzier R, Lesieur B, Werkoff G, Antoine M, Rodenas A, Darai E, Chereau E. Expression of somatostatin type-2 and -4 receptor and correlation with histological type in breast cancer. Anticancer Res. 2014 Aug;34(8):3997-4003. PMID 25075022
- [Background] Dude I, Zhang Z, Rousseau J, Hundal-Jabal N, Colpo N, Merkens H, Lin KS, Benard F. Evaluation of agonist and antagonist radioligands for somatostatin receptor imaging of breast cancer using positron emission tomography. EJNMMI Radiopharm Chem. 2017;2(1):4. doi: 10.1186/s41181-017-0023-y. Epub 2017 Apr 17. PMID 29503845
- [Background] Sollini M, Erba PA, Fraternali A, Casali M, Di Paolo ML, Froio A, Frasoldati A, Versari A. PET and PET/CT with 68gallium-labeled somatostatin analogues in Non GEP-NETs Tumors. ScientificWorldJournal. 2014 Feb 13;2014:194123. doi: 10.1155/2014/194123. eCollection 2014. PMID 24693229
- [Background] Dalm SU, Haeck J, Doeswijk GN, de Blois E, de Jong M, van Deurzen CHM. SSTR-Mediated Imaging in Breast Cancer: Is There a Role for Radiolabeled Somatostatin Receptor Antagonists? J Nucl Med. 2017 Oct;58(10):1609-1614. doi: 10.2967/jnumed.116.189035. Epub 2017 Apr 27. PMID 28450563
- [Background] Dalm SU, Schrijver WA, Sieuwerts AM, Look MP, Ziel-van der Made AC, de Weerd V, Martens JW, van Diest PJ, de Jong M, van Deurzen CH. Prospects of Targeting the Gastrin Releasing Peptide Receptor and Somatostatin Receptor 2 for Nuclear Imaging and Therapy in Metastatic Breast Cancer. PLoS One. 2017 Jan 20;12(1):e0170536. doi: 10.1371/journal.pone.0170536. eCollection 2017. PMID 28107508
- [Background] Hope TA, Bergsland EK, Bozkurt MF, Graham M, Heaney AP, Herrmann K, Howe JR, Kulke MH, Kunz PL, Mailman J, May L, Metz DC, Millo C, O'Dorisio S, Reidy-Lagunes DL, Soulen MC, Strosberg JR. Appropriate Use Criteria for Somatostatin Receptor PET Imaging in Neuroendocrine Tumors. J Nucl Med. 2018 Jan;59(1):66-74. doi: 10.2967/jnumed.117.202275. Epub 2017 Oct 12. No abstract available. PMID 29025982
- [Background] Ozelius L, Kramer PL, Moskowitz CB, Kwiatkowski DJ, Brin MF, Bressman SB, Schuback DE, Falk CT, Risch N, de Leon D, et al. Human gene for torsion dystonia located on chromosome 9q32-q34. Neuron. 1989 May;2(5):1427-34. doi: 10.1016/0896-6273(89)90188-8. PMID 2576373
- [Background] Virgolini I, Ambrosini V, Bomanji JB, Baum RP, Fanti S, Gabriel M, Papathanasiou ND, Pepe G, Oyen W, De Cristoforo C, Chiti A. Procedure guidelines for PET/CT tumour imaging with 68Ga-DOTA-conjugated peptides: 68Ga-DOTA-TOC, 68Ga-DOTA-NOC, 68Ga-DOTA-TATE. Eur J Nucl Med Mol Imaging. 2010 Oct;37(10):2004-10. doi: 10.1007/s00259-010-1512-3. PMID 20596866
- See also: Fiche info - SOMAKIT TOC 40 microgrammes, trousse pour préparation radiopharmaceutique - Base de données publique des médicaments. — https://base-donnees-publique.medicaments.gouv.fr/extrait.php?specid=65028549
- See also: 111In-Pentetreotide Scintigraphy Versus 68Ga-DOTATATE PET: Impact on Krenning Scores and Effect of Tumor Burden — http://www.google.com/search?client=firefox-b-1-d&q=111In-Pentetreotide+Scintigraphy+Versus+68Ga-